CLINICAL TRIAL: NCT06892002
Title: A Real-World Observational Study Characterizing Patients With Type 1 Diabetes Treated With Teplizumab
Brief Title: Description of Patients With Type 1 Diabetes Treated With Teplizumab
Acronym: TEPLI-REAL
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: PDE0109; U1111-1315-4417 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-01-24; First posted 2025-03-24 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
Keywords: Teplizumab; Type 1 Diabetes; Real-world study; Stage 2 Type 1 Diabetes; Stage 3 Type 1 Diabetes; Disease progression; Treatment patterns; Patient monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Disease Progression | interventions — teplizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Teplizumab treated participants: Participants who received teplizumab as part of their routine clinical care
  Interventions: Drug: Teplizumab

INTERVENTIONS:
Drug: Teplizumab — This study will not administer any treatment, only observe the treatment as prescribed in real-world clinical practice.

SUMMARY:
Type 1 diabetes mellitus (T1D) is a chronic autoimmune disease caused by the destruction of pancreatic β cells. T1D pathogenesis progresses through several stages: Stage 1 T1D includes the presence of β cell autoimmunity and thus presence of islet autoantibodies, without the presence of dysglycemia and symptoms. Stage 2 T1D includes the presence of islet autoantibodies and dysglycemia, also with no symptoms. Stage 3 T1D includes presence of islet autoantibodies, overt hyperglycemia, and symptoms; most patients with Stage 3 T1D meet standard diagnostic criteria for diabetes and require insulin treatment.

Teplizumab has been shown to delay progression to Stage 3 in participants at Stage 2 in a Phase 2 clinical trial, leading to subsequent approval in the United States of America (USA). Patients outside of the USA are able to receive the treatment through Pre-Registration Import Licenses and Managed Access Programs. The current study will collect data on the use of teplizumab in routine care, to better understand which patients received teplizumab and how these patients were managed after they received the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient informed consent or assent (for patients < 18 years old) according to local regulations or appropriate informed consent waivers prior to any study related activity.
* Patient received ≥ 1 day of teplizumab treatment.

Exclusion Criteria:

* Participation in an interventional clinical study on the index date. Participation in an interventional clinical study is defined as initiating the product/procedure or control under investigation. An interventional clinical study is a study that requires deviation from standard clinical practice by following a study protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients whose index date (teplizumab initiation date) was ≥ 6 weeks before site activation and who meet the eligibility criteria outlined below will be eligible for enrollment into the study.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Participant demographic characteristics at teplizumab initiation | At Day 1 (first dose of teplizumab)
  Age, sex at birth, race (for US participants only), ethnicity (for US participants only), height, weight, Body mass index (BMI)
Participants' family history of T1D and autoimmune diseases | At Day 1 (first dose of teplizumab)
  First- and second-degree relatives with T1D
Presence of T1D susceptibility genes: Genetic risk score | At Day 1 (first dose of teplizumab)
Presence of T1D susceptibility genes: Human Leukocyte Antigen (HLA)-haplotype | At Day 1 (first dose of teplizumab)
Participants' medical history | From 6 months prior to the first dose of teplizumab (teplizumab initiation) (or the earliest date of all data contributing to Stage 2 T1D diagnosis, whichever is earlier) up to the medical records abstraction date, approximately 3-4 years
  Date of stage 1 confirmation, date of dysglycemia confirmation
Assessment of blood glucose test results: CGM | At screening (6 months before teplizumab initiation), within 6 weeks prior to teplizumab initiation, during teplizumab infusion (2 weeks), following completion of teplizumab treatment (through study completion, up to 30 months)"

SECONDARY OUTCOMES:
Development of stages of T1D | From the date of first assessment of dysglycemia or positive autoantibody test up to date of first dose of teplizumab (teplizumab initiation), approximately 6 months to 1 year
  Patient monitoring for T1D progression from early to late stages
Assessment of blood glucose test results: HbA1c | At screening (6 months before teplizumab initiation), within 6 weeks prior to teplizumab initiation, during teplizumab infusion (2 weeks), following completion of teplizumab treatment (through study completion, up to 30 months)"
Assessment of blood glucose test results: Fasting Plasma Glucose (FPG) | At screening (6 months before teplizumab initiation), within 6 weeks prior to teplizumab initiation, during teplizumab infusion (2 weeks), following completion of teplizumab treatment (through study completion, up to 30 months)"
Assessment of blood glucose: Oral glucose tolerance test (OGTT) | At screening (6 months before teplizumab initiation), within 6 weeks prior to teplizumab initiation, during teplizumab infusion (2 weeks), following completion of teplizumab treatment (through study completion, up to 30 months)"
Assessment of blood glucose test results: Random Plasma Glucose (PG) | At screening (6 months before teplizumab initiation), within 6 weeks prior to teplizumab initiation, during teplizumab infusion (2 weeks), following completion of teplizumab treatment (through study completion, up to 30 months)"
Assessment of bloog glucose test results: Continuous glucose monitoring (CGM) | At screening (6 months before teplizumab initiation), within 6 weeks prior to teplizumab initiation, during teplizumab infusion (2 weeks), following completion of teplizumab treatment (through study completion, up to 30 months)"
Assessment of blood glucose test results: Post-prandial glucose (PPG) | At screening (6 months before teplizumab initiation), within 6 weeks prior to teplizumab initiation, during teplizumab infusion (2 weeks), following completion of teplizumab treatment (through study completion, up to 30 months)"
Assessment of autoantibody tests results | At screening (6 months before teplizumab initiation), within 6 weeks prior to teplizumab initiation, during teplizumab infusion (2 weeks), following completion of teplizumab treatment (through study completion, up to 30 months)"
  Anti-GAD65, IAA, Anti-IA-2, ICA, Anti-ZnT8
Assessment of C-peptide test results | At screening (6 months before teplizumab initiation), within 6 weeks prior to teplizumab initiation, during teplizumab infusion (2 weeks), following completion of teplizumab treatment (through study completion, up to 30 months)"
Treatments participants received: teplizumab treatment and other treatments | From earliest of 6 months or the earliest date of all data contributing to Stage 2 T1D diagnosis (i.e. first record of dysglycemia and/or positive autoantibody test) and after teplizumab treatment until end of follow-up, approximately 3-4 years
  Teplizumab treatment and other treatment variables (insulin, other glucose lowering agents)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (24):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - University of California, San Francisco, San Francisco, California
  - Barbara Davis Center For Childhood Diabetes, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami Medical Center, Miami, Florida
  - USF Diabetes Center, Tampa, Florida
  - Doctor's Clinic, Vero Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Riley Hospital for Children, Carmel, Indiana
  - University of Louisville, Louisville, Kentucky
  - Boston Children's Hospital Division of Endocrinology, Boston, Massachusetts
  - Atlantic Health, Morristown, New Jersey
  - Hassenfeld Children's Hospital at NYU Langone, New York, New York
  - Morgan Stanley Children's Hospital, New York, New York
  - Ten's Medical PC, Staten Island, New York
  - SUNY Upstate Medical University PARENT, Syracuse, New York
  - Sanford Research/USD, Fargo, North Dakota
  - AM Diabetes & Endocrinology Center, Bartlett, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - El Paso Medical Research Institute, El Paso, Texas
  - University of Utah Hospitals & Clinics, Salt Lake City, Utah
  - Diabetes and Endocrine Treatment Specialists, Sandy City, Utah
- Israel (3):
  - Schneider Children's Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org